CLINICAL TRIAL: NCT02342834
Title: Mechanisms Through Which a Small Protein and Lipid Preload Improves Glucose Tolerance in Subjects With Impaired Glucose Homeostasis
Brief Title: Effects of a Small Protein and Lipid Preload on Glucose Tolerance in Subjects With Impaired Glucose Homeostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Andrea Natali, Professor, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LISBONA
Record Dates: First submitted 2015-01-13; First posted 2015-01-21 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): During the "control" study, each subject ingest 500 ml of water 30 minutes before a standard 75 g Oral Glucose Tolerance Test
- Small mixed protein and lipid meal (Experimental): During the "preload" study, each subject ingest a small mixed meal 30 minutes before a standard 75 g Oral Glucose Tolerance Test. The meal is composed by 50 g of parmesan cheese, one small size boiled egg and 300 ml of water (250 kcal, 23 g protein, 17 g fat and 2 g of carbohydrate).
  Interventions: Dietary Supplement: Small mixed protein and lipid meal

INTERVENTIONS:
Dietary Supplement: Small mixed protein and lipid meal — Ingestion of a small mixed protein and lipid meal 30 minutes before glucose
  Arms: Small mixed protein and lipid meal

SUMMARY:
The purpose of this study is:

* to measure the size of the effect on glucose tolerance of a small mixed protein and lipid meal given as a pre-load in individuals with different glucose tolerance status
* to investigate the underlying mechanisms by accurately evaluating beta cell function, insulin sensitivity, insulin clearance and glucose kinetics (oral absorption, endogenous production, rate of utilization) together with gut hormones plasma concentration.

DETAILED DESCRIPTION:
As supported by experimental and clinical data, oral carbohydrate tolerance is influenced by the coingestion of nutrients through multiple mechanisms. The ingestion itself, the contact with the gastric mucosa, the arrival into the intestine and the subsequent digestion are known to produce neural reflexes, hormonal responses and plasma substrates gradients which, by modulating gastric emptying, insulin secretion and insulin clearance participate in the regulation of postprandial glycaemia. The size of this effect is influenced by a number of factors: the specific nutrient chemical characteristics (fat vs protein and composition) and their physical properties (solid vs liquid), the timing (pre-load vs coingestion) and finally the individual glucose tolerance status. To our knowledge, the effect on glucose excursions of a combination of protein and fat given before carbohydrate is still unknown and also unknown is the contribution of different mechanisms involved in the control of glucose homeostasis in subjects with different degrees of glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* healthy, prediabetic or diet-controlled type 2 diabetic patients
* Subjects ≥ 18 and ≤65 years of age
* Lean, Overweight or Obese (BMI: 18 to 35 kg/m2)
* Normal liver and kidney function
* Normal thyroid function
* Read and understood the informed consent form and signed it voluntarily

Exclusion Criteria:

* Liver, heart, kidney, lung, infectious, neurological, psychiatric, immunological or neoplastic diseases.
* Type 1 or insulin treated diabetes.
* Pregnancy or lactation
* Illicit drug abuse or alcoholism
* Subject treated with insulin or treatment
* Subjects taking anoretic drugs
* Subjects on steroid treatment
* Subjects after bariatric surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-01; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Plasma glucose response during the Oral Glucose Tolerance Test | 120 minutes

SECONDARY OUTCOMES:
Insulin secretion, estimated from C-peptide deconvolution | 120 minutes
Insulin sensitivity, estimated from glucose and insulin levels during the Oral Glucose Tolerance Test with the use of Oral Glucose Insulin Sensitivity index | 120 minutes
  The Oral Glucose Insulin Sensitivity index (OGIS; equation for a 2-h oral glucose test with a glucose dose of 75 g) is the mean glucose clearance change (basal vs OGTT 60-120 min), divided by the mean plasma insulin concentration gradient over the same time interval.
Insulin clearance, estimated by calculating the Insulin secretion/Plasma insulin ratio | 120 minutes
Glucose fluxes (intestinal glucose absorption, endogenous glucose production, rate of disappearance of plasma glucose), assessed by modeling glucose tracers enrichments using a standard double tracers technique | 120 minutes
Incretin secretion (plasma GLP-1, plasma GIP) | 120 minutes
Plasma glucagon | 120 minutes
Plasma Non Esterified Fatty Acids | 120 minutes
Beta cells function parameters (glucose sensitivity, rate sensitivity, potentiation factor ratio), calculated by modeling insulin secretion and glucose concentration. | 120 minutes
Endothelial function assessed as the reactive hyperemia index by an EndoPAT device | fasting, 60 min and 120 min during the control and preload OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natali, Professor, Study Chair — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy

REFERENCES:
- [Derived] Trico D, Frascerra S, Baldi S, Mengozzi A, Nesti L, Mari A, Natali A. The insulinotropic effect of a high-protein nutrient preload is mediated by the increase of plasma amino acids in type 2 diabetes. Eur J Nutr. 2019 Sep;58(6):2253-2261. doi: 10.1007/s00394-018-1778-y. Epub 2018 Jul 14. PMID 30008106
- [Derived] Trico D, Baldi S, Tulipani A, Frascerra S, Macedo MP, Mari A, Ferrannini E, Natali A. Mechanisms through which a small protein and lipid preload improves glucose tolerance. Diabetologia. 2015 Nov;58(11):2503-12. doi: 10.1007/s00125-015-3710-9. Epub 2015 Jul 30. PMID 26224101